CLINICAL TRIAL: NCT06864169
Title: A Phase 2 Nonrandomized, Open-label, Multisite Study to Evaluate the Safety and Efficacy of Raludotatug Deruxtecan in Participants With Gastrointestinal Cancers
Brief Title: A Study of Raludotatug Deruxtecan (R-DXd) in People With Gastrointestinal Cancers (MK-5909-005)
Acronym: REJOICE-GI01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5909-005; 2024-517416-30-00 (Other: EU CT); U1111-1312-2472 (Other: UTN)
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Raludotatug Deruxtecan (R-DXd) (Experimental): R-DXd will be administered via IV infusion.
  Interventions: Biological: Raludotatug Deruxtecan (R-DXd)

INTERVENTIONS:
Biological: Raludotatug Deruxtecan (R-DXd) — Administered via intravenous (IV) infusion.
  Other Names: MK-5909; DS 6000a

SUMMARY:
Researchers are looking for new ways to treat certain types of advanced gastrointestinal (GI) cancers. The study medicine raludotatug deruxtecan (also called MK-5909, R-DXd, or DS-6000a) is a type of medicine called an antibody-drug conjugate (ADC). An ADC attaches to a protein on cancer cells and delivers treatment to destroy those cells.

The main goal of this study is to learn if the cancer responds to treatment (gets smaller or goes away).

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has one of the following cancers:

  * Unresectable or metastatic pancreatic ductal adenocarcinoma (PDAC)
  * Unresectable or metastatic adenocarcinoma of the biliary tract [intra- or extrahepatic holangiocarcinoma (CCA) or gallbladder cancer (GBC)]
  * Unresectable or metastatic colorectal adenocarcinoma
  * Unresectable or metastatic gastric adenocarcinoma
  * Gastroesophageal junction adenocarcinoma (GEJAC)
  * Esophageal adenocarcinoma (EAC)
* Has received prior therapy for the cancer
* Has a life expectancy of at least 3 months
* If human immunodeficiency virus (HIV) infected, must have well controlled HIV on antiretroviral therapy (ART)

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a history of (noninfectious) interstitial lung disease (ILD)/pneumonitis that required steroids or has current ILD/pneumonitis, and/or suspected ILD/pneumonitis
* Has clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses
* Has uncontrolled or significant cardiovascular disease
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in the past 2 years
* Has not adequately recovered from major surgery or has ongoing surgical complications
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-07-06 (Estimated); Study Completion 2029-01-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 15 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience CR or PR as assessed by BICR will be presented.

SECONDARY OUTCOMES:
Number of Participants who Experience One or More Adverse Events (AEs) | Up to approximately 14 months
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants who Discontinue Study Treatment due to an AE | Up to approximately 12 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.
Duration of Response (DOR) | Up to approximately 49 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Progression Free Survival (PFS) | Up to approximately 49 months
  PFS is defined as the time from first day of study intervention to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by BICR. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 49 months
  OS is defined as the time from the first dose to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (41):
- United States (8):
  - Yale New Haven Hospital ( Site 0375), New Haven, Connecticut
  - Sibley Memorial Hospital ( Site 0372), Washington D.C., District of Columbia
  - Mt Sinai Comprehensive Cancer Center ( Site 0345), Miami Beach, Florida
  - St. Vincent Healthcare Frontier Cancer Center ( Site 0347), Billings, Montana
  - Morristown Medical Center ( Site 0349), Morristown, New Jersey
  - University Hospitals Cleveland Medical Center ( Site 0369), Cleveland, Ohio
  - University of Virginia Cancer Center ( Site 0365), Charlottesville, Virginia
  - University of Wisconsin Carbone Cancer Center ( Site 0348), Madison, Wisconsin
- Argentina (4):
  - Instituto de Investigaciones Clinicas Mar del Plata ( Site 0001), Mar del Plata, Buenos Aires
  - Nefra Medical Care - CEMIC Saavedra ( Site 0008), Buenos Aires, Buenos Aires F.D.
  - Instituto Medico de la Fundacion Estudios Clinicos ( Site 0007), Rosario, Santa Fe Province
  - Fundación CORI para la Investigación y Prevención del Cáncer ( Site 0006), La Rioja
- Canada (3):
  - Sunnybrook Research Institute ( Site 0044), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0041), Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal ( Site 0042), Montreal, Quebec
- Chile (4):
  - FALP ( Site 0062), Santiago, Region M. de Santiago
  - Centro de Estudios Clínicos SAGA ( Site 0064), Santiago, Region M. de Santiago
  - Clínica UC San Carlos de Apoquindo ( Site 0066), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0069), Santiago, Region M. de Santiago
- France (4):
  - Centre François Baclesse ( Site 0085), Caen, Calvados
  - Institut Regional du Cancer Montpellier ( Site 0084), Montpellier, Herault
  - Pitie Salpetriere University Hospital ( Site 0082), Paris, Orne
  - Gustave Roussy ( Site 0081), Villejuif, Val-de-Marne
- Hong Kong (2):
  - Prince of Wales Hospital ( Site 0122), Hksar
  - Queen Mary Hospital ( Site 0121), Hksar
- Spain (5):
  - Institut Català d'Oncologia (ICO) - Badalona ( Site 0222), Badalona, Barcelona
  - Hospital Universitario Marqués de Valdecilla ( Site 0221), Santander, Cantabria
  - Hospital Clinic de Barcelona ( Site 0223), Barcelona
  - Hospital General Universitario Gregorio Marañón ( Site 0225), Madrid
  - Hospital Universitario Fundacion Jimenez Diaz ( Site 0224), Madrid
- Switzerland (3):
  - Universitaetsspital Basel ( Site 0241), Basel, Canton of Basel-City
  - Hôpitaux Universitaires de Genève (HUG) ( Site 0245), Geneva, Canton of Geneva
  - Universitaetsspital Zuerich ( Site 0242), Zurich
- Taiwan (6):
  - China Medical University Hospital ( Site 0267), Taichung
  - Taichung Veterans General Hospital ( Site 0265), Taichung
  - National Cheng Kung University Hospital ( Site 0263), Tainan
  - National Taiwan University Hospital ( Site 0261), Taipei
  - Mackay Memorial Hospital ( Site 0266), Taipei
  - Taipei Veterans General Hospital ( Site 0262), Taipei
- Thailand (2):
  - Ramathibodi Hospital. ( Site 0282), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 0281), Bangkok, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com